CLINICAL TRIAL: NCT01086410
Title: Study HZA106851: A Study of the Effects of Inhaled Fluticasone Furoate/GW642444 Versus Placebo on the HPA Axis of Adolescent and Adult Asthmatics
Brief Title: Safety Study of the Effects of Inhaled Fluticasone Furoate/GW642444 on the Hypothalamic-Pituitary-Adrenal (HPA) Axis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106851
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: HPA axis
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- FF/444 Dose B (Active Comparator): Fluticasone furoate/GW642444 Dose B inhalation powder once daily for 6 weeks' treatment + 1 oral placebo capsule each day on the last 7 days of the study
  Interventions: Drug: Fluticasone Furoate/GW642444 Inhalation Powder; Drug: Placebo Oral Capsule
- FF/444 Dose A (Active Comparator): Fluticasone furoate/GW642444 Dose A inhalation powder once daily for 6 weeks' treatment + 1 oral placebo capsule each day on the last 7 days of the study
  Interventions: Drug: Fluticasone Furoate/GW642444 Inhalation Powder; Drug: Placebo Oral Capsule
- Placebo (Placebo Comparator): Placebo inhalation powder once daily for 6 weeks' treatment + 1 oral placebo capsule each day on the last 7 days of the study
  Interventions: Drug: Placebo Inhalation Powder; Drug: Placebo Oral Capsule
- Prednisolone (Active Comparator): Placebo inhalation powder once daily for 6 weeks' treatment + 1 oral prednisolone 10mg capsule each day on the last 7 days of the study
  Interventions: Drug: Placebo Inhalation Powder; Drug: Prednisolone Oral Capsule

INTERVENTIONS:
Drug: Placebo Inhalation Powder — Placebo Inhalation powder inhaled once daily for 6 weeks' treatment
  Arms: Placebo; Prednisolone
Drug: Fluticasone Furoate/GW642444 Inhalation Powder — Dose B inhaled once daily for 6 weeks' treatment
  Arms: FF/444 Dose B
Drug: Fluticasone Furoate/GW642444 Inhalation Powder — Dose A inhaled once daily for 6 weeks' treatment
  Arms: FF/444 Dose A
Drug: Placebo Oral Capsule — One placebo capsule taken each day on the last 7 days of the study
  Arms: FF/444 Dose A; FF/444 Dose B; Placebo
Drug: Prednisolone Oral Capsule — Prednisolone 10mg oral capsule taken each day on the last 7 days of the study
  Arms: Prednisolone

SUMMARY:
The purpose of this study is to assess the effect of six weeks' treatment with two once-daily strengths of Fluticasone Furoate/GW642444 Inhalation Powder on the HPA axis system

ELIGIBILITY:
Inclusion Criteria:

* Outpatient with ability to comply with study requirements and complete two 24-hour clinic visits
* Clinical diagnosis of asthma for greater than/equal to 12 weeks
* Reversibility FEV1 of at least twelve percent and two hundred milliliters
* FEV1 greater than or equal to fifty percent of predicted

Exclusion Criteria:

* History of life threatening asthma
* Respiratory infection or oral candidiasis
* Asthma exacerbation
* Uncontrolled disease or clinical abnormality
* Allergies to study drugs, study drugs' excipients, medications related to study drugs
* Taking another investigational medication or prohibited medication

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (4):
  - GSK Investigational Site, Cypress, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, San Antonio, Texas
- Germany (5):
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Poland (7):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gidle
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 106851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the inclusion criteria entered a 7- to 14-day Run-in Period (screening visit [Visit 1]). Participants were provided with albuterol/salbutamol inhalation aerosol for relief of asthma symptoms during the study.
Pre-assignment Details: At the end of the Run-in Period, participants who meet the randomization criteria were admitted to the clinic in the evening (Visit 2) for the Baseline collection of 24-hour serial serum cortisol samples and urine. Eligible participants were randomly assigned to one of four treatment groups in a 4:4:4:1 ratio.
Groups:
- Placebo: Participants received placebo via a Dry Powder Inhaler (DPI) for 6 weeks, plus a placebo capsule on the last 7 days of treatment. Participants were instructed to self-administer one inhalation from the DPI once daily at approximately the same time each evening for 6 weeks and to take one placebo capsule each morning on the last 7 days of treatment.
- FF/VI 100/25 µg PM: Participants received Fluticasone Furoate/Vilanterol (FF/VI) 100/25 micrograms (µg) via a DPI for 6 weeks, plus a placebo capsule on the last 7 days of treatment. Participants were instructed to self-administer one inhalation from the DPI once daily at approximately the same time each evening (PM) for 6 weeks and to take one placebo capsule each morning (AM) on the last 7 days of treatment.
- FF/VI 200/25 µg PM: Participants received FF/VI 200/25 µg via a DPI for 6 weeks, plus a placebo capsule on the last 7 days of treatment. Participants were instructed to self-administer one inhalation from the DPI once daily at approximately the same time each evening (PM) for 6 weeks and to take one placebo capsule each morning (AM) on the last 7 days of treatment.
- Prednisolone 10 mg AM: Participants received placebo via a DPI for 6 weeks, plus a prednisolone 10 milligram (mg) capsule on the last 7 days of treatment. Participants were instructed to self-administer one inhalation of placebo from the DPI once daily at approximately the same time each evening (PM) for 6 weeks and to take one Prednisolone capsule each morning (AM) on the last 7 days of treatment.
Period: Overall Study
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Started | 58 | 56 | 56 | 15
Completed | 55 | 54 | 55 | 13
Not Completed | 3 | 2 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 2
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM | Total
Number analyzed (Participants) | 58 | 56 | 56 | 15 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (15.42) | 34.4 (15.63) | 34.0 (13.74) | 37.5 (14.19) | 35.1 (14.82)
Gender [Count of Participants; unit: Participants]
  Female | 27 | 31 | 23 | 6 | 87
  Male | 31 | 25 | 33 | 9 | 98
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3 | 0 | 1 | 0 | 4
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian - Japanese Heritage | 0 | 0 | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 55 | 56 | 53 | 15 | 179

OUTCOME MEASURES:

1. Primary Outcome: Ratio From Baseline of the Serum Cortisol Weighted Mean (0-24 Hours) on Day -1/1 (Baseline) and Day 42
Description: Serum cortisol weighted mean was determined for each participant over the time period 0-12 hours on Day -1/1 (Baseline) and Day 42. Serum cortisol weighted mean was derived by dividing the area under the concentration-time curve (AUC; defined as thearea under the concentration-time curve from time zero up to 24 hours) by the sample collection time interval. The sample collection time interval is defined as the difference between the time of the last cortisol sample and the time of the first cortisol sample. Samples were collected at the following time points: 0 (first blood draw/pre-dose); 2, 4, 9, 12, 14, 16, 20, 22, and 24 hours (relative to the "0" time point). Because values are on a logged scale, the ratio of the endpoint to Baseline is presented, as it is a measure of the difference from Baseline.
Time Frame: Day -1/1 (Baseline) and Day 42
Population: Serum Cortisol (SC) Population: all participants in the Intent-to-Treat Population who did not have protocol deviations that were considered to affect the SC endpoint and whose serum samples were not considered to have confounding factors affecting results interpretation. Only those participant available at the specified time points were analzyed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio from Baseline
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 52 | 50 | 53 | 13
ratio from Baseline | 0.99 (29.6) | 0.99 (40.0) | 0.96 (27.2) | 0.32 (72.9)
Statistical Analysis 1: Comparison: Placebo vs FF/VI 100/25 µg PM; Test type: Superiority or Other; Ratio of least square gometric mean = 0.99, 95% CI 2-sided [0.87 to 1.12] — Analysis was performed using Analysis of Covariance (ANCOVA) with covariates of region, sex, age, treatment, and the log of the Baseline values
Statistical Analysis 2: Comparison: Placebo vs FF/VI 200/25 µg PM; Test type: Superiority or Other; Ratio of least square gometric mean = 0.97, 95% CI 2-sided [0.86 to 1.10] — Analysis was performed using ANCOVA with covariates of region, sex, age, treatment, and the log of the Baseline values
Statistical Analysis 3: Comparison: Placebo vs Prednisolone 10 mg AM; Test type: Superiority or Other; Ratio of least square gometric mean = 0.34, 95% CI 2-sided [0.28 to 0.41] — Analysis performed using ANCOVA with covariates of region, sex, age, treatment, and the log of the Baseline values

2. Secondary Outcome: Ratio From Baseline of the Serum Cortisol Area Under the Concentration-time Curve (AUC) (0-24 Hour) on Day -1/1 (Baseline) and Day 42
Description: Area under the plasma drug concentration-time (AUC[0-24 hour]) curve from time zero (pre-dose) to the last time of quantifiable serum cortisol concentration at 24 hours post-dose on Day -1/1 (Baseline) and Day 42 was measured. AUC reflects the actual body exposure to drug over a specified period of time after administration of a dose. Samples were collected at the following times: 0 (immediately pre-dose inhaled study drug); post-dose at 5 minutes (min), 15 min, 30 min, and 1 hour (hr), 2 hr, 4 hr, 9 hr, 12 hr, 16 hr, 20 hr, and 24 hr. Because values are on a logged scale, the ratio of the endpoint to Baseline is presented, as it is a measure of the difference from Baseline.
Time Frame: Day -1/1 (Baseline) and Day 42
Population: SC Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio from Baseline
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 52 | 50 | 53 | 13
ratio from Baseline | 0.99 (29.6) | 0.99 (40.1) | 0.97 (27.2) | 0.32 (71.9)

3. Secondary Outcome: Ratio From Baseline of Serum Cortisol Trough (0-24 Hours) at Day -1/1 (Baseline) and Day 42
Description: Serum cortisol trough is defined as the minimum value of serum cortisol measured over the 24-hour period. Samples were collected at the following times: 0 (immediately pre-dose inhaled study drug); post-dose at 5 minutes (min), 15 min, 30 min, and 1 hour (hr), 2 hr, 4 hr, 9 hr, 12 hr, 16 hr, 20 hr, and 24 hr. Because values are on a logged scale, the ratio of the endpoint to Baseline is presented, as it is a measure of the difference from Baseline.
Time Frame: Day -1/1 (Baseline) and Day 42
Population: SC Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio from Baseline
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 52 | 51 | 53 | 13
ratio from Baseline | 1.04 (88.2) | 0.84 (88.7) | 0.73 (80.7) | 0.28 (82.3)

4. Secondary Outcome: Ratio From Baseline of 0-24 Hour Urinary Free Cortisol Excretion on Day -1/1 (Baseline) and Day 42
Description: A 24-hour urine sample was collected for the measurement of 24-hour urinary cortisol excretion at Day -1/1 (Baseline) and Day 42. Only those participants available at the specified time points were analyzed. Because values are on a logged scale, the ratio of the endpoint to Baseline is presented, as it is a measure of the difference from Baseline.
Time Frame: Day -1/1 (Baseline) and Day 42
Population: Urine Cortisol (UC) Population: all participants in the ITT Population who did not have protocol deviations that were considered to affect the urine cortisol endpoint and whose urine samples were not considered to have confounding factors that would affect the interpretation of the results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio from Baseline
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 49 | 47 | 53 | 12
ratio from Baseline | 0.87 (77.923) | 1.03 (110.952) | 0.92 (96.312) | 0.40 (204.433)

5. Secondary Outcome: Plasma FF and VI Pharmacokinetic (PK) Concentration
Description: Plasma FF and VI Pharmacokinetic (PK) Concentration were estimates at the following time points:0 (immediately pre-dose inhaled study drug), and post-dose at 5 min, 15 min, 30 min, and 1 hr, 2 hr, 4 hr, 9 hr, 12 hr, 16 hr, 20 hr, 24 hr on Day 42. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the Pharmacokinetic Population.
Time Frame: Day 42
Population: Pharmacokinetic (PK) Population: all participants in the ITT Population for whom a pharmacokinetic sample was obtained and analyzed.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 0 | 54 | 56 | 0
picograms per milliliter (pg/mL)
  FF, 0 hour, n=53, 54 |  | 3.57 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 10.02 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  FF, 5 minutes post-dose, n=51, 54 |  | 16.65 (10.191) | 25.55 (14.438) |
  FF, 15 minutes post-dose, n=50, 54 |  | 16.35 (10.198) | 28.84 (14.441) |
  FF, 30 minutes post-dose, n=52, 52 |  | 17.12 (10.583) | 30.68 (15.461) |
  FF, 1 hour post-dose, n=54, 54 |  | 16.91 (9.637) | 30.07 (15.540) |
  FF, 2 hours post-dose, n=51, 53 |  | 15.00 (9.272) | 30.20 (18.292) |
  FF, 4 hours post-dose, n=54, 53 |  | 9.78 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 21.79 (11.597) |
  FF, 9 hours post-dose, n=48, 52 |  | 6.20 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 15.99 (11.667) |
  FF, 12 hours post-dose, n=51, 55 |  | 4.62 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 13.37 (9.670) |
  FF, 16 hours post-dose, n=49, 52 |  | 2.55 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 11.73 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  FF, 20 hours post-dose, n=51, 51 |  | 1.74 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 9.28 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  FF, 24 hours post-dose, n=48, 53 |  | 1.55 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 7.58 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  VI, 0 hours, n=52, 54 |  | 2.57 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 7.95 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  VI, 5 minutes post-dose, n=50, 54 |  | 85.22 (70.582) | 90.54 (88.794) |
  VI, 15 minutes post-dose, n=48, 55 |  | 62.94 (52.020) | 72.53 (55.271) |
  VI, 30 minutes post-dose, n=51, 55 |  | 33.38 (33.932) | 36.88 (33.157) |
  VI, 1 hour post-dose, n=52, 53 |  | 14.63 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 20.07 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  VI, 2 hours post-dose, n=52, 55 |  | 7.09 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 6.06 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  VI, 4 hours post-dose, n=52, 54 |  | 0.00 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 0.45 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  VI, 9 hours post-dose, n=52, 55 |  | 0.00 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 0.47 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  VI, 12 hours post-dose, n=52, 55 |  | 0.00 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 1.21 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  VI, 16 hours post-dose, n=51, 52 |  | 0.00 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 4.76 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  VI, 20 hours post-dose, n=50, 54 |  | 0.00 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 0.00 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |
  VI, 24 hours post-dose, n=52, 55 |  | 1.19 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. | 0.00 (NA) — Values below 10 pg/mL are below the limit of quantification and are imputed. Standard deviation is not displayed if >30% of values are imputed. |

6. Secondary Outcome: AUC(0-t) and AUC(0-24) for FF on Day 42
Description: Area under the plasma drug concentration-time (AUC[0-t]) curve from time zero (pre-dose) to the last time of quantifiable FF concentration and AUC(0-24) is the concentration time curve from zero (pre-dose) to 24 hours of quantifiable FF concentration on Day 42 was measured. AUC reflects the actual body exposure to drug over a specified period of time after administration of a dose. Samples were collected at the following times: 0 (immediately pre-dose inhaled study drug); post-dose at 5 minutes (min), 15 min, 30 min, and 1 hour (hr), 2 hr, 4 hr, 9 hr, 12 hr, 16 hr, 20 hr, and 24 hr post-dose on Day 42.
Time Frame: Day 42
Population: PK Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the PK Population.
Measure: Geometric Mean (95% Confidence Interval); unit: picograms*hour per milliliter (pg*hr/mL)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 0 | 54 | 56 | 0
picograms*hour per milliliter (pg*hr/mL)
  AUC(0-t), n=54, 55 |  | 58.842 [37.706 to 91.825] | 221.694 [152.697 to 321.868] |
  AUC(0-24), n=49, 53 |  | NA [NA to NA] — Data are not available because >=50% of values were non-calculable due to non-quantifiable concentrations (below the level of detection). | 324.015 [267.233 to 392.862] |

7. Secondary Outcome: Cmax for FF on Day 42
Description: Cmax is defined as the maximum observed concentration on Day 42. Samples were collected at the following times: 0 (immediately pre-dose inhaled study drug); post-dose at 5 minutes (min), 15 min, 30 min, and 1 hour (hr), 2 hr, 4 hr, 9 hr, 12 hr, 16 hr, 20 hr, and 24 hr post-dose on Day 42.
Time Frame: Day 42
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 0 | 54 | 55 | 0
picograms per milliliter (pg/mL) |  | 19.388 [16.796 to 22.379] | 33.017 [28.586 to 38.135] |

8. Secondary Outcome: Tmax and Tlast of FF at Day 42
Description: tmax is defined as the time to reach the observed maximum concentration, and tlast is defined as the time of the last observed quantifiable concentration on Day 42. Samples were collected at the following times: 0 (immediately pre-dose inhaled study drug); post-dose at 5 minutes (min), 15 min, 30 min, and 1hour (hr), 2 hr, 4 hr, 9 hr, 12 hr, 16 hr, 20 hr, and 24 hr post-dose on Day 42.
Time Frame: Day 42
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 0 | 54 | 55 | 0
hours
  tmax |  | 0.500 [0.03 to 8.97] | 0.500 [0.07 to 4.00] |
  tlast |  | 9.000 [0.98 to 24.00] | 20.042 [0.95 to 24.08] |

9. Secondary Outcome: AUC(0-t) for VI on Day 42
Description: Area under the concentration-time (AUC[0-t]) curve from time zero (pre-dose) to the last time of quantifiable VI concentration on Day 42 was measured. Samples were collected at the following times: 0 (immediately pre-dose inhaled study drug); post-dose at 5 minutes (min), 15 min, 30 min, and 1 hour (hr), 2 hr, 4 hr, 9 hr, 12 hr, 16 hr, 20 hr, and 24 hr post-dose on Day 42.
Time Frame: Day 42
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: picograms*hour per milliliter (pg*hr/mL)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 0 | 52 | 55 | 0
picograms*hour per milliliter (pg*hr/mL) |  | 41.177 (53.9720) | 66.937 (142.3461) |

10. Secondary Outcome: Cmax for VI on Day 42
Description: as for outcome 7
Time Frame: Day 42
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 0 | 52 | 55 | 0
picograms per milliliter (pg/mL) |  | 101.227 (73.8233) | 118.531 (86.8659) |

11. Secondary Outcome: Tmax and Tlast of VI at Day 42
Description: tmax is defined as the time to reach the observed maximum concentration, and tlast is defined as the time of the last observed quantifiable VI concentration on Day 42. Samples were collected at the following times: 0 (immediately pre-dose inhaled study drug); post-dose at 5 minutes (min), 15 min, 30 min, and 1hour (hr), 2 hr, 4 hr, 9 hr, 12 hr, 16 hr, 20 hr, and 24 hr post-dose on Day 42.
Time Frame: Day 42
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 0 | 52 | 55 | 0
hours
  tmax |  | 0.083 [0.00 to 2.00] | 0.083 [0.00 to 16.00] |
  tlast |  | 0.500 [0.03 to 2.00] | 0.950 [0.08 to 16.00] |

12. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations. Refer to the General Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the start of study medication until Day 42 (Visit 5)/Early Withdrawal
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
Participants
  Any AE | 16 | 23 | 21 | 5
  Any SAE | 0 | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in Basophil, Eosinophil, Lymphocyte, Monocyte, and Segmented Neutrophil Values at Day 42/Early Withdrawal (EW)
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, and segmented neutrophils at Baseline and Day 42/EW. For all laboratory assessments, Baseline is the most recent recorded value at Screening or prior to Day -1/1. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value.
Time Frame: Baseline and Day 42/Early Withdrawal (EW)
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
Percentage
  Basophils, Day 42, n=50, 47, 53, 11 | 0.05 (0.354) | 0.04 (0.356) | -0.05 (0.350) | -0.08 (0.223)
  Basophils, EW, n=2, 2, 0, 0 | -0.10 (0.141) | 0.10 (0.141) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Eosinophils, Day 42, n=50, 47, 53, 11 | 0.57 (2.837) | 0.27 (2.073) | -0.99 (2.664) | -1.11 (1.488)
  Eosinophils, EW, n=2, 2, 0, 0 | 0.50 (0.849) | -0.55 (2.051) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Lymphocytes, Day 42, n=50, 47, 53, 11 | 1.09 (6.836) | 1.54 (8.853) | -1.32 (7.844) | -2.48 (14.319)
  Lymphocytes, EW, n=2, 2, 0, 0 | 2.90 (10.607) | 2.00 (2.263) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Monocytes, Day 42, n=50, 47, 53, 11 | -0.51 (2.074) | -0.03 (3.333) | 0.07 (2.581) | -0.70 (1.977)
  Monocytes, EW, n=2, 2, 0, 0 | -1.00 (0.424) | -0.70 (3.111) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Segmented Neutrophils, Day 42, n=50, 47, 53, 11 | -1.16 (8.291) | -1.85 (10.279) | 2.30 (9.583) | 4.37 (15.667)
  Segmented Neutrophils, EW, n=2, 2, 0, 0 | -2.30 (11.738) | -0.85 (3.465) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.

14. Secondary Outcome: Change From Baseline in Eosinophil, Total Neutrophil, Platelet, and White Blood Cell (WBC) Count Values at Day 42/EW
Description: Blood samples were collected for the measurement of eosinophils, total neutrophils, platelets, and WBC count at Baseline and Day 42/EW. For all laboratory assessments, Baseline is the most recent recorded value at Screening or prior to Day -1/1. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value.
Time Frame: Baseline and Day 42/EW
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
10^9 cells per liter (GI/L)
  Eosinophils, Day 42, n=50, 47, 53, 11 | 0.066 (0.2282) | 0.044 (0.1608) | -0.022 (0.1805) | -0.036 (0.0803)
  Eosinophils, EW, n=2, 2, 0, 0 | 0.015 (0.0071) | -0.060 (0.1697) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Total Neutrophils, Day 42, n=50, 47, 53, 11 | 0.017 (1.3317) | 0.289 (1.4873) | 0.704 (1.2403) | 1.435 (2.5515)
  Total Neutrophils, EW, n=2, 2, 0, 0 | -0.420 (1.7253) | -1.165 (0.9970) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Platelets, Day 42, n=50, 48, 51, 11 | -11.1 (28.72) | -8.2 (31.33) | -3.9 (25.31) | 16.1 (16.50)
  Platelets, EW, n=1, 2, 0, 0 | -2.0 (NA) — Data are not available (missing) for some participants who withdrew from the study early. | -39.5 (28.99) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  WBC Day 42, n=50, 47, 53, 11 | 0.22 (1.584) | 0.71 (1.787) | 0.96 (1.367) | 1.69 (2.418)
  WBC EW, n=2, 2 | -0.25 (1.344) | -1.65 (0.778) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.

15. Secondary Outcome: Change From Baseline in Hemoglobin Values at Day 42/EW
Description: Blood samples were collected for the measurement of hemoglobin at Baseline and Day 42/EW. For all laboratory assessments, Baseline is the most recent recorded value at Screening or prior to Day -1/1. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value.
Time Frame: Baseline and Day 42/EW
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
Grams per liter (g/L)
  Day 42, n=50, 48, 53, 11 | -5.8 (10.28) | -6.2 (6.23) | -5.7 (6.59) | -3.5 (9.27)
  EW, n=2, 2, 0, 0 | -10.5 (2.12) | -3.0 (8.49) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.

16. Secondary Outcome: Change From Baseline in Hematocrit Values at Day 42/EW
Description: Blood samples were collected for the measurement of hematocrit at Baseline and Day 42/EW. For all laboratory assessments, Baseline is the most recent recorded value at Screening or prior to Day -1/1. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value.
Time Frame: Baseline and Day 42/EW
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Proportion of 1
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
Proportion of 1
  Day 42, n=50, 48, 53, 11 | -0.0123 (0.02957) | -0.0120 (0.02125) | -0.0114 (0.02151) | -0.0072 (0.02955)
  EW, n=2, 2, 0, 0 | -0.0175 (0.00071) | -0.0050 (0.02263) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.

17. Secondary Outcome: Change From Baseline in Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Creatine Kinase (CK), and Gamma Glutamyl Transferase (GGT) Values at Day 42/EW
Description: Blood samples were collected for the measurement of ALT, ALP, AST, CK, and GGT at Baseline and Day 42/EW. For all laboratory assessments, Baseline is the most recent recorded value at Screening or prior to Day -1/1. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value.
Time Frame: Baseline and Day 42/EW
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
International units per liter (IU/L)
  ALT, Day 42, n=55, 51, 55, 12 | -1.3 (13.05) | -2.0 (8.49) | -2.2 (10.86) | 0.8 (3.33)
  ALT, EW, n=2, 2, 0, 0 | -5.0 (8.49) | 0.5 (2.12) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  ALP, Day 42, n=55, 51, 55, 12 | -6.8 (11.06) | -2.1 (13.96) | -2.6 (8.33) | -4.9 (9.86)
  ALP, EW, n=2, 2, 0, 0 | 1.5 (9.19) | -1.0 (1.41) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  AST, Day 42, n=54, 50, 51, 12 | -0.1 (12.42) | -1.4 (6.82) | -0.6 (6.91) | -1.8 (5.67)
  AST, EW, n=2, 2, 0, 0 | 0.5 (0.71) | 0.0 (1.41) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  CK, Day 42, n=55, 51, 55, 12 | -42.3 (342.74) | -18.5 (289.98) | 5.5 (67.57) | -17.3 (95.02)
  CK, EW, n=2, 2, 0, 0 | 15.0 (21.21) | 33.0 (73.54) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  GGT, Day 42, n=55, 51, 55, 12 | -3.3 (10.65) | -2.5 (6.94) | 2.2 (17.24) | 3.1 (7.32)
  GGT, EW, n=2, 2, 0, 0 | -2.5 (6.36) | -0.5 (0.71) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.

18. Secondary Outcome: Change From Baseline in Albumin and Total Protein Values at Day 42/EW
Description: Blood samples were collected for the measurement of albumin and total protein at Baseline and Day 42/EW. For all laboratory assessments, Baseline is the most recent recorded value at Screening or prior to Day -1/1. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value.
Time Frame: Baseline and Day 42/EW
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
Grams per liter
  Albumin, Day 42, n=55, 51, 55, 12 | -2.7 (3.29) | -1.5 (3.02) | -1.3 (3.11) | -0.3 (2.81)
  Albumin, EW, n=2, 2, 0, 0 | -1.5 (3.54) | 0.5 (2.12) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Total Protein, Day 42, n=55, 51, 55, 12 | -4.1 (5.06) | -1.9 (4.39) | -1.8 (4.65) | -0.8 (4.18)
  Total Protein, EW, n=2, 2, 0, 0 | -0.5 (3.54) | 0.0 (0.00) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.

19. Secondary Outcome: Change From Baseline in Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, and Creatinine Values at Day 42/EW
Description: Blood samples were collected for the measurement of direct bilirubin, indirect bilirubin, total bilirubin, and creatinine at Baseline and Day 42/EW. For all laboratory assessments, Baseline is the most recent recorded value at Screening or prior to Day -1/1. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value.
Time Frame: Baseline and Day 42/EW
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
Micromoles per liter (µmol/L)
  Direct Bilirubin, Day 42, n=55, 51, 55, 12 | -0.6 (1.12) | -0.6 (1.02) | -0.5 (1.10) | 0.3 (0.75)
  Direct Bilirubin, EW, n=2, 2, 0, 0 | -1.0 (0.00) | 0.0 (0.00) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Indirect Bilirubin, Day 42, n=55, 51, 55, 12 | -2.0 (4.89) | -2.5 (3.20) | -1.4 (4.72) | -1.0 (2.76)
  Indirect Bilirubin, EW, n=2, 2, 0, 0 | -1.5 (2.12) | -2.0 (0.00) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Total Bilirubin, Day 42, n=55, 51, 55, 12 | -2.5 (5.66) | -3.2 (3.72) | -1.8 (5.67) | -0.8 (2.86)
  Total Bilirubin, EW, n=2, 2, 0, 0 | -2.5 (2.12) | -2.0 (0.00) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Creatinine, Day 42, n=55, 51, 55, 12 | -0.41 (8.688) | 0.35 (8.088) | 0.04 (8.052) | 4.61 (9.585)
  Creatinine, EW, n=2, 2, 0, 0 | 0.00 (13.435) | 0.95 (6.435) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.

20. Secondary Outcome: Change From Baseline in Chloride, Carbon Dioxide (CO2) Content/Bicarbonate, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) Values at Day 42/EW
Description: Blood samples were collected for the measurement of chloride, carbon dioxide (CO2) content/bicarbonate, glucose, potassium, sodium, and urea/blood urea nitrogen (BUN) at Baseline and Day 42/EW. For all laboratory assessments, Baseline is the most recent recorded value at Screening or prior to Day -1/1. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value.
Time Frame: Baseline and Day 42/EW
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
Millimoles per liter (mmol/L)
  Chloride, Day 42, n=55, 51, 55, 12 | 1.2 (2.54) | 0.9 (2.76) | 0.7 (3.06) | -1.0 (2.41)
  Chloride, EW, n=2, 2, 0, 0 | 2.0 (1.41) | -0.5 (0.71) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  CO2 content/bicarbonate, Day 42, n=54, 50, 51, 12 | -1.0 (2.86) | -2.0 (2.98) | -1.5 (2.35) | -0.1 (3.12)
  CO2 content/bicarbonate, EW, n=2, 2, 0, 0 | -3.5 (2.12) | 0.0 (1.41) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Glucose, Day 42, n=55, 51, 55, 12 | 0.11 (1.117) | 0.23 (1.037) | -0.03 (0.573) | 0.40 (1.397)
  Glucose, EW, n=2, 2, 0, 0 | 1.00 (0.283) | 0.40 (0.849) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Potassium, Day 42, n=54, 50, 51, 12 | -0.10 (0.385) | -0.11 (0.405) | -0.16 (0.379) | 0.03 (0.599)
  Potassium, EW, n=2, 2, 0, 0 | -0.20 (0.283) | -0.65 (0.071) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Sodium, Day 42, n=55, 51, 55, 12 | 0.0 (2.03) | -0.1 (1.98) | -0.1 (3.01) | -0.2 (1.85)
  Sodium, EW, n=2, 2, 0, 0 | 1.5 (3.54) | -3.5 (0.71) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.
  Urea/BUN, Day 42, n=55, 51, 55, 12 | -0.14 (1.432) | 0.48 (1.441) | -0.00 (1.236) | 0.94 (1.331)
  Urea/BUN, EW, n=2, 2, 0, 0 | 1.30 (0.283) | -0.85 (0.919) | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early. | NA (NA) — Data are not available (missing) for some participants who withdrew from the study early.

21. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Days 14, 28, 42, and Maximum Post-Baseline
Description: SBP and DBP were measured at Baseline and at Days 14, 28, 42, and EW. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value. Scheduled, unscheduled, and early withdrawal visits were used for the maximum post-Baseline assessment.
Time Frame: Days 14, 28, 42, and EW
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
Millimeters of mercury (mmHg)
  SBP, Day 14, n=58, 55, 56, 14 | -0.5 (11.68) | -1.9 (10.88) | -1.3 (10.53) | -1.0 (13.33)
  SBP, Day 28, n=57, 55, 56, 14 | -0.9 (9.55) | -0.7 (10.70) | -2.3 (11.66) | -3.9 (13.35)
  SBP, Day 42, n=55, 54, 56, 13 | 2.3 (11.96) | -0.4 (12.72) | -1.8 (11.20) | 1.5 (8.26)
  SBP, maximum post-Baseline, n=58, 56, 56, 15 | 6.2 (11.44) | 5.0 (10.88) | 3.9 (10.80) | 4.9 (8.61)
  DBP, Day 14, n=58, 55, 56, 14 | 0.0 (7.92) | -1.1 (8.26) | -0.6 (9.08) | 0.1 (8.55)
  DBP, Day 28, n=57, 55, 56, 14 | 1.8 (8.38) | -0.6 (7.63) | 0.1 (9.97) | -0.4 (8.11)
  DBP, Day 42, n=55, 54, 56, 13 | 1.2 (8.77) | -1.2 (9.13) | 0.3 (8.74) | 1.2 (8.69)
  DBP, maximum post-Baseline, n=58, 56, 56, 15 | -3.3 (7.04) | -5.2 (7.76) | -5.4 (9.00) | -4.9 (7.97)

22. Secondary Outcome: Change From Baseline in Pulse Rate at Days 14, 28, 42, and Maximum Post-Baseline
Description: Heart rate was measured at Baseline and at Days 14, 28, 42, and EW. Change from Baseline was calculated as the Day 42/EW value minus the Baseline value. Scheduled, unscheduled, and early withdrawal visits were used for the maximum post-Baseline assessment.
Time Frame: Days 14, 28, 42, and EW
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Number analyzed (Participants) | 58 | 56 | 56 | 15
Beats per minute
  Day 14, n=58, 55, 56, 14 | 1.5 (13.05) | 1.7 (10.70) | 0.0 (8.72) | -1.8 (7.92)
  Day 28, n=57, 55, 56, 14 | 2.9 (13.45) | -0.9 (9.32) | -1.9 (12.05) | -2.7 (11.89)
  Day 42, n=55, 54, 56, 13 | -0.1 (12.65) | -0.9 (11.43) | 0.9 (8.96) | -2.3 (9.10)
  Maximum post-Baseline, n=58, 56, 56, 15 | 8.0 (12.47) | 6.0 (9.86) | 5.5 (8.64) | 2.9 (9.13)

ADVERSE EVENTS:
Arm/Group | Placebo | FF/VI 100/25 µg PM | FF/VI 200/25 µg PM | Prednisolone 10 mg AM
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/56 | 0/56 | 0/15
Other Adverse Events (participants affected / at risk) | 9/58 | 20/56 | 13/56 | 5/15
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=58) | FF/VI 100/25 µg PM (N=56) | FF/VI 200/25 µg PM (N=56) | Prednisolone 10 mg AM (N=15)
Headache (Nervous system disorders) | 5 | 15 | 9 | 2
Sinus headache (Nervous system disorders) | 0 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Facial palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.